CLINICAL TRIAL: NCT05364073
Title: A Phase 1b Dose Escalation and Dose Expansion Study Evaluating the Safety, Pharmacokinetics, and Antitumor Activity of Furmonertinib in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Activating Epidermal Growth Factor Receptor (EGFR) or Human Epidermal Growth Factor Receptor 2 (HER2) Mutations
Brief Title: Study of Furmonertinib in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Activating, Including Uncommon, Epidermal Growth Factor Receptor (EGFR) or Human Epidermal Growth Factor Receptor 2 (HER2) Mutations
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ArriVent BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FURMO-002
Record Dates: First submitted 2022-04-06; First posted 2022-05-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Metastatic Non-Small Cell Lung Cancer; Advanced Non-Small Cell Lung Cancer; HER2 Exon 20 Mutations; EGFR Exon 20 Mutations; EGFR Uncommon Mutations, Including G719X and S768I
Keywords: Non-small cell lung cancer (NSCLC); Metastatic Non-Small Cell Lung Cancer; Advanced Non-Small Cell Lung Cancer; EGFR; HER2; Exon 20 Insertion Mutations; HER2 kinase domain mutations; Epidermal Growth Factor Receptor (EGFR) kinase domain mutations; Exon 20; Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Mutations; HER2 Exon 20 Insertion Mutations; Tyrosine Kinase Inhibitor (TKI); Human Epidermal Growth Factor Receptor 2 (HER2); Epidermal Growth Factor Receptor (EGFR); EGFR uncommon mutations; EGFR atypical mutations; EGFR rare mutations; V774M; G719X; S768I; E709X; R776C/H; G724S; E736K; I740_K745dup; N771G; K757M/R; V769L/M; T854X; T751_I759delinsN; G719A; G719S; R776C; R776H; K757M; K757R; V769L; V769M; osimertinib; afatinib; E709_T710del insD; G779F; L747X
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1 Dose Escalation and Backfill (Experimental): Experimental: Previously treated patients with advanced or metastatic NSCLC with activating EGFR or HER2 mutations
  Interventions: Drug: Furmonertinib
- Stage 2 Expansion Cohort 1 (Experimental): Previously Treated NSCLC Patients with EGFR Exon 20 Insertion Mutations
  Interventions: Drug: Furmonertinib
- Stage 2 Expansion Cohort 2 (Experimental): Previously treated NSCLC Patients with HER2 Exon 20 Insertion Mutations
  Interventions: Drug: Furmonertinib
- Stage 2 Expansion Cohort 3 (Experimental): Previously treated NSCLC Patients with EGFR Activating Mutations, who are not eligible for Cohorts 1 and 4
  Interventions: Drug: Furmonertinib
- Stage 2 Expansion Cohort 4 (Experimental): Untreated or Previously treated EGFR TKI Naïve NSCLC Patients with EGFR Uncommon Mutations, excluding EGFR exon 20 insertion mutations
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib tablet
  Other Names: AST2818
  Arms: Stage 1 Dose Escalation and Backfill
Drug: Furmonertinib — Furmonertinib tablet
  Other Names: AST2818
  Arms: Stage 2 Expansion Cohort 1
Drug: Furmonertinib — Furmonertinib tablet
  Other Names: AST2818
  Arms: Stage 2 Expansion Cohort 2
Drug: Furmonertinib — Furmonertinib tablet
  Other Names: AST2818
  Arms: Stage 2 Expansion Cohort 3
Drug: Furmonertinib — Furmonertinib tablet
  Other Names: AST2818
  Arms: Stage 2 Expansion Cohort 4

SUMMARY:
This is a Phase 1b, open-label, multi-center, dose-escalation and dose expansion study designed to evaluate the safety, pharmacokinetics (PK), and preliminary antitumor activity of furmonertinib in patients with advanced or metastatic non-small cell lung cancer (NSCLC) with activating, including uncommon, Epidermal Growth Factor Receptor (EGFR) or Human Epidermal Growth Factor Receptor 2 (HER2) mutations. Patients will be enrolled into one of 2 stages: Stage 1 (Dose Escalation and Backfill Cohorts) and Stage 2 (Dose Expansion).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) not amenable to curative surgery or radiotherapy.
* Disease that has progressed after at least one available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable; or for whom a clinical trial of an investigational agent is a recognized standard of care.
* Documented radiologic disease progression during or after the last systemic anti-cancer therapy before the first dose of furmonertinib.
* For patients with Epidermal Growth Factor Receptor (EGFR) mutations sensitive to osimertinib, the patient must have received osimertinib prior to study enrollment in regions where osimertinib is approved, including the US.

Stage 1 dose escalation and backfill cohorts and Stage 2 Cohorts 1, 2, 3 and 4:

-Patients with CNS metastases (including leptomeningeal disease) may be eligible if meeting additional protocol specified criteria.

Stage 1 Dose Escalation and Backfill Cohorts Inclusion Criteria:

- Documented validated results from local testing of tumor tissue or blood confirming the presence of an activating, including uncommon, EGFR mutation or HER2 exon 20 insertion mutation performed at a CLIA-or equivalently certified laboratory.

Stage 2 Cohort 1 Previously Treated, Locally Advanced or Metastatic NSCLC Patients with EGFR Exon 20 Insertion Mutations Inclusion Criteria

* Documented validated results from local testing of either tumor tissue or blood confirming the presence of EGFR Exon 20 insertion mutations, performed at a CLIA- or equivalently certified laboratory.
* The patient must have experienced disease progression or have intolerance to treatment with platinum-based chemotherapy.

Stage 2 Cohort 2 Previously treated, Locally Advanced or Metastatic NSCLC Patients with HER2 Exon 20 Insertion Mutations Inclusion Criteria

* Documented validated results from local testing of either tumor tissue or blood confirming the presence of HER2 Exon 20 insertion mutations, performed at a CLIA- or equivalently certified laboratory.
* The patient must have experienced disease progression or have intolerance to treatment with platinum-based chemotherapy.
* In regions in which fam-trastuzumab deruxtecan-nxki is approved and available for adult patients with unresectable or metastatic NSCLC whose tumors have activating HER2 exon 20 mutations, the patient must have received or be considered not appropriate to receive fam-trastuzumab deruxtecan-nxki.

Stage 2 Cohort 3 Previously Treated, Locally Advanced or Metastatic NSCLC Patients with EGFR Activating Mutations Mutations, who are not eligible for Cohorts 1 and 4 Inclusion Criteria

* Documented validated results from local testing of either tumor tissue or blood confirming the presence of an EGFR activating mutation, performed at a CLIA- or equivalently certified laboratory.
* The patient must have experienced disease progression or have intolerance to treatment with the standard of care EGFR TKI.
* Patients with CNS metastases may be eligible if meeting additional protocol specified criteria.

Stage 2 Cohort 4 Untreated or Previously Treated EGFR TKI-Naïve, Locally Advanced or Metastatic NSCLC Patients with EGFR Uncommon Mutations excluding EGFR Exon 20 insertions Inclusion Criteria

* Previously untreated in the locally advanced or metastatic setting or have progressed after at least 1 available standard therapy, or for whom standard therapy has proven to be ineffective, intolerable, or considered inappropriate
* Documented validated results from local testing of either tumor tissue or blood confirming the presence of an EGFR Uncommon mutation, performed at a CLIA- or equivalently certified laboratory a. Representative mutations include, but are not limited to, G719X, S768I, E709X, G779F, L747X, V774M, E709_T710delinsD, R776C/H, G724S, E736K, I740_K745dup, N771G, K757M/R, V769L/M, T854X, T751_I759delinsN

Key Exclusion Criteria:

* Treatment with chemotherapy, targeted therapy, biologic therapy or an investigational agent as anti-cancer therapy within 3 or 3 elimination weeks or five half-lives prior to initiation of furmonertinib, whichever is shorter, or endocrine therapy within 2 weeks prior to initiation of furmonertinib.
* Radiation therapy as cancer therapy within 4 weeks prior to initiation of furmonertinib.
* Palliative radiation to bone metastases within 2 weeks prior to initiation of furmonertinib.
* AE from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia or Grade ≤ 2 peripheral neuropathy.

Stage 2 Cohort 4 Untreated or Previously Treated EGFR TKI-Naïve, Locally Advanced or Metastatic NSCLC Patients with EGFR Uncommon Mutations Exclusion Criteria

* Prior treatment with any EGFR TKIs
* Progression during neoadjuvant or adjuvant therapy (e.g., chemotherapy, radiotherapy, immunotherapy or investigational agents) or within 12 months of completion of above therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Number of incidence and severity of adverse events (AEs) as a measure of safety and tolerability of Furmonertinib | Up to 36 months after first dose
Stage 2: Overall Response Rate (ORR) | Up to 36 months after first dose

SECONDARY OUTCOMES:
Stage 1: Overall Response Rate | Up to 36 months after first dose
Stage 1: Duration of Response (DOR) | Up to 36 months after first dose
Stage 1: Disease Control Rate | Up to 36 months after first dose
Stage 1: Progression Free Survival | Up to 36 months after first dose
Stage 1: Depth of Response | Up to 36 months after first dose
Stage 1: Overall survival | Up to 36 months after first dose
Stage 1: Central Nervous System ORR | Up to 36 months after first dose
Stage 1: Central Nervous System DOR | Up to 36 months after first dose
Stage 1: Plasma concentrations of furmonertinib and its major metabolite (AST5902) | Up to 36 months after first dose
Stage 1, Cohort 1, Backfill only: Plasma concentrations of furmonertinib and its major metabolite (AST5902) | Up to 36 months after first dose
Stage 1, Cohort 1, Backfill only: Plasma concentrations of midazolam and its metabolite (1-OH-midazolam) | Up to 36 months after first dose
Stage 2, all cohorts: Duration of Response | Up to 36 months after first dose
Stage 2, all cohorts: Disease Control Rate | Up to 36 months after first dose
Stage 2, all cohorts: Progression Free Survival | Up to 36 months after first dose
Stage 2, all cohorts: Depth of Response | Up to 36 months after first dose
Stage 2, all cohorts: Overall survival | Up to 36 months after first dose
Stage 2, all cohorts: Central Nervous System ORR | Up to 36 months after first dose
Stage 2, all cohorts: Central Nervous System DOR | Up to 36 months after first dose
Stage 2, Cohort 4 only: Overall Response Rate | Up to 36 months after first dose
Stage 2, all cohorts: Number of incidence and severity of AEs as a measure of safety and tolerability of Furmonertinib | Up to 36 months after first dose
Stage 2, all cohorts: Plasma concentrations of furmonertinib and its major metabolite (AST5902) | Up to 36 months after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Lam, Study Director — ArriVent BioPharma
Locations (39):
- United States (7):
  - ArriVent Investigative Site, Prescott, Arizona
  - ArriVent Investigative Site, Sacramento, California
  - ArriVent Investigative Site, Whittier, California
  - ArriVent Investigative Site, Celebration, Florida
  - ArriVent Investigative Site, Detroit, Michigan
  - ArriVent Investigative Site, Houston, Texas
  - ArriVent Investigative Site, Fairfax, Virginia
- Australia (3):
  - ArriVent Investigative Site, Blacktown, New South Wales
  - ArriVent Investigative Site, St Leonards, New South Wales
  - ArriVent Investigative Site, Heidelberg, Victoria
- Canada (2):
  - Arrivent Investigative Site, Edmonton
  - Arrivent Investigative Site, Toronto
- China (12):
  - Allist Investigative Site, Hefei, Anhui
  - Allist Investigative Site, Beijing, Beijing Municipality
  - Allist Investigative Site, Chaoyang, Beijing Municipality
  - Allist Investigative Site, Chongqing, Chongqing Municipality
  - Allist Investigative Site, Harbin, Heilongjiang
  - Allist Investigative Site, Zhengzhou, Henan
  - Allist Investigative Site, Wuhan, Hubei
  - Allist Investigative Site, Xuzhou, Jiangsu
  - Allist Investigative Site, Nanchang, Jianxi
  - Allist Investigative Site, Changchun, Jilin
  - Allist Investigative Site, Jinan, Shandong
  - Allist Investigative Site, Taiyuan, Shanxi
- France (3):
  - ArriVent Investigative Site, Lyon
  - Arrivent Investigative Site, Toulouse
  - Arrivent Investigative Site, Villejuif
- ArriVent Investigative Site, Medolla, Italy
- Japan (4):
  - ArriVent Investigative Site, Chiba, Chiba
  - Arrivent Investigative Site, Ōsaka-sayama, Osaka
  - Arrivent Investigative Site, Chūō, Tokyo
  - Arrivent Investigative Site, Koto-Ku, Tokyo
- Arrivent Investigative Site, Amsterdam, North Holland, Netherlands
- South Korea (2):
  - Arrivent Investigative Site, Gwangju
  - Arrivent Investigative Site, Seoul
- Spain (3):
  - ArriVent Investigative Site, Barcelona
  - ArriVent Investigative Site, Madrid
  - ArriVent Investigative Site, Valencia
- ArriVent Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No